CLINICAL TRIAL: NCT06756438
Title: Efficacy Evaluation and Cutaneous Acceptibility of a Dermocosmetic Product on Subjects Suffering of Atopic Dermatisis - Study Vs Placebo -- Use Test Under Dermatological Control -
Brief Title: Efficacy Evaluation and Cutaneous Acceptibility of a Dermocosmetic Product on Subjects Suffering of Atopic Dermatisis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NAOS Les Laboratoires (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC2024PSaib+PL
Record Dates: First submitted 2024-11-28; First posted 2025-01-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: ATOPIC DERMATITIS; Eczema; Dermocosmetic
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: This study was conducted under a double-blind, randomized, multicenter, before-and-after, parallel-group design. Participants received either the test product or a placebo, while continuing topical corticosteroid treatment in combination or as a relay.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amr 1: Study product (Experimental): Product 1: Study product, Emollient. Face and body
  Interventions: Other: Study product
- Arm 2: Placebo (Placebo Comparator): Product 2: Placebo, Emollient. face and body
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Study product — Anti-itching, anti-replapse and repairing treatment. Emollient.
  Arms: Amr 1: Study product
Other: Placebo — Emollient
  Arms: Arm 2: Placebo

SUMMARY:
Atopic eczema is a chronic inflammatory skin disease, mainly affecting children, characterized by itching and flare-ups. It results from genetic and environmental factors, leading to immunological and cutaneous abnormalities.

The aim of this study is to assess the efficacy of a product for atopic skin versus a placebo. Primary objectives include assessing the number, the delay and severity of recurrences of atopic dermatitis (measured by the SCORAD score), and the evolution of symptoms such as dryness and pruritus. Secondary objectives include quality of life and quality of sleep and skin acceptability.

The study protocol is a multicenter, double-blind, randomized clinical trial, in which participants receive either the study product or a placebo, while continuing their topical corticosteroid treatment.

ELIGIBILITY:
Inclusion Criteria:

Specific

* Sex: female and/or male;
* Age: from 3 months up to 12 years old;
* Phototype: I to IV;
* 100% with atopic skin;
* 100% with sensitive skin;
* Subject who had at least 3 eczema flares-up of atopic dermatitis during the last 6 months before start of the study, including the crisis observed on D-X.
* Subject presenting on the visit D-X a flare-up of eczema for which the dermatologist prescribed treatment with topical corticosteroids treatment;
* Subjects with SCORAD between 15 and 40 on D-X;
* Subject who do not require medical treatment anymore after using prescribed topical corticosteroids from D-X up to D0 and clinical signs of atopic dermatitis are resolved, to be defined on D0 visit (in case of insufficient healing of inflammatory lesions, the subject continues medical treatment as recommended by the investigator).

General

* Healthy subject;
* Child whose at least one parent/legal guardian has given freely and expressly her/his informed consent;
* Child whose at least one parent/legal guardian is willing to adhere to the protocol and study procedures;
* Polish citizenship.

Exclusion Criteria:

* Cutaneous pathology on the study zone other than atopic dermatitis;
* Use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the efficacy of the study products, including anti-histaminic treatment (except prescribed dermocorticoids on D-X and in case of flare-up during the study course);
* Subject having undergone a surgery under general anesthesia within the previous month;
* Excessive exposure to sunlight or UV-rays within the previous month;
* Subject enrolled in another clinical trial during the study period (concerns the studied zones);
* Subjects presenting oozing eczema lesions or any sign of infection on eczema lesions (e.g; pus).

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
SCOring Atopic Dermatisis (SCORAD) | Before (Day-X) and after the products use (Day 0, Month 2, Month 4 and Month 6)
  The SCORAD (Scoring Atopic Dermatitis) scale ranges from a minimum score of 0 to a maximum score of 103, where higher scores indicate a worse outcome, reflecting more severe atopic dermatitis.
SCORING ATOPIC DERMATITIS BY SUBJECT'S PARENT/LEGAL GUARDIAN (PO-SCORAD) | Before (Day -X) and after the products use (Day 0, Month 2, Month 4 and Month 6)
  The PO-SCORAD ( Patient-Oriented SCOring Atopid Dermatisis) scale ranges from a minimum score of 0 to a maximum score of 75, where higher scores indicate a worse outcome, reflecting more severe atopic dermatitis.
CUTANEOUS ACEPTABILITY | On Day 0, Month 2, Month 4 and Month 6 of the product use, the body and face of the subject is examined by the dermatologist in charge of the study.
  The product's capacity to maintain human body in good condition (cutaneous acceptability) by clinical examination by the dermatologist in charge of the study to assess each following parameters : erythema, edema, dryness, desquamation, roughness, fonctional and physical signs.
Evaluation of "xerosis", "pruritus" and "insomnia" evolution based on SCORAD | Before (Day-X) and after the products use (Day 0, Month 2, Month 4 and Month 6)
  The SCORAD (Scoring Atopic Dermatitis) scale ranges from a minimum score of 0 to a maximum score of 103, where higher scores indicate a worse outcome, reflecting more severe atopic dermatitis.

CONTACTS AND LOCATIONS:
Locations (1):
- EUROFINS, Gdansk, Poméranie, Poland

IPD SHARING:
Plan to Share IPD: No